CLINICAL TRIAL: NCT04022629
Title: Acute Shoulder Stabilisation Using Endoscopic Techniques (ASSET) 2 Study: Long-Term Follow-up of a Randomised Control Trial
Brief Title: ASSET 2 Study: Long-Term Follow-up of a Randomised Control Trial
Acronym: ASSET 2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royal Infirmary of Edinburgh (Other)
Responsible Party: Principal Investigator, Liam Yapp, Specialty Registrar, Royal Infirmary of Edinburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC19020
Record Dates: First submitted 2019-07-07; First posted 2019-07-17 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group 1 (Active Comparator): Patients aged between 18-35 years who have sustained a first-time traumatic anterior dislocation of the shoulder.
  Interventions: Procedure: Arthroscopic Washout Only
- Treatment Group 2 (Active Comparator): Patients aged between 18-35 years who have sustained a first-time traumatic anterior dislocation of the shoulder.
  Interventions: Procedure: Arthroscopic Bankart Repair

INTERVENTIONS:
Procedure: Arthroscopic Washout Only — To wash out the shoulder joint with a sterile solution through an arthroscope (keyhole surgery) under a general anaesthetic.
  Arms: Treatment Group 1
Procedure: Arthroscopic Bankart Repair — To repair the torn glenoid labrum in the shoulder, using key-hole (arthroscopic) surgery techniques under general anaesthetic. The Bankart technique is well described and will be performed using suture anchors.
  Arms: Treatment Group 2

SUMMARY:
This study aims to measure the long-term efficacy of arthroscopic Bankart repair for first-time anterior shoulder dislocation in terms of recurrent instability and functional outcome.

DETAILED DESCRIPTION:
Approximately half of patients who experience a dislocation of their shoulder will go on to experience further problems with their shoulder. Some people will suffer persisting instability, and notice an uncomfortable feeling of their shoulder wanting to give way. This can occur commonly during active movements such as playing sports or lifting heavy objects. Some patients experience recurrent dislocations, and find that their shoulder is so weak that it slips out of joint with little provocation.

Previous research suggested that this high rate of subsequent shoulder problems can be greatly reduced (although not abolished completely) by surgery performed soon after the first dislocation. Ten years ago, there were two different methods which had been popularised:

1. Arthroscopic Wash-Out: The first is to wash out the shoulder joint with a sterile solution through an arthroscope (keyhole surgery) under a general anaesthetic.
2. Arthroscopic Repair: The second is to repair the torn tissues in the shoulder, again using key-hole surgery techniques under general anaesthetic.

A previous clinical trial was undertaken in our unit (2001-2005) which randomised young patients aged under 35 years to one of the two possible treatments (described above). These procedures were not new or experimental. The same Arthroscopic Repair technique continues to be routinely used in NHS Lothian to treat patients who have late problems following a dislocated shoulder. We do not routinely perform wash-outs of the shoulder joint because this is only effective in treating problems that occur at an early stage.This new study intends to build on these findings by asking each of the patient groups to complete a short questionnaire which uses validated outcomes to measure their shoulder function. The aim of the study is to identify if there is a long-term clinical and functional benefit of early arthroscopic shoulder stabilisation in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients who had previously enrolled in the previous study shall be considered eligible for inclusion.
* Aged between 25 and 55 years.

Exclusion Criteria:

* Patients will be excluded from this long-term follow-up if no contact details are available or if they no longer retained the capacity to provide consent to participate in the study

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Recurrent Dislocation | Up to 20 years post-surgery
  Radiographic evidence of recurrent dislocation

SECONDARY OUTCOMES:
Disabilities of Shoulder, elbow and Hand (DASH) scores | Up to 20 years post-surgery
  Objective validated measure of general upper limb function. Comparison between pre-operative, 2 year post-operative and long-term (10-20 year) post-operative total score of each cohort. Score calculated to give a total out of 100. The lower the score, the better the function.
Western Ontario Shoulder Instability (WOSI) Index. | Up to 20 years post-surgery
  Objective validated measure of instability-specific shoulder function. Comparison between pre-operative, 2 year post-operative and long-term (10-20 year) post-operative total score of each cohort. Total score is out of 2100.

CONTACTS AND LOCATIONS:
Overall Officials: Liam Z Yapp, MRCSEd, Principal Investigator — NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No patient identifiable data shall be available to anyone other than the study researchers.

REFERENCES:
- [Background] Robinson CM, Jenkins PJ, White TO, Ker A, Will E. Primary arthroscopic stabilization for a first-time anterior dislocation of the shoulder. A randomized, double-blind trial. J Bone Joint Surg Am. 2008 Apr;90(4):708-21. doi: 10.2106/JBJS.G.00679. PMID 18381306